CLINICAL TRIAL: NCT07303972
Title: Electrical Impedance Tomography Saline Indicator Technique for Assessing Differences in Lung Perfusion Between Inspiratory and Expiratory Breath-Hold Phases: A Prospective Self-Controlled Study
Brief Title: Effects of Inspiratory vs Expiratory Breath-Hold on Lung Perfusion Measured by EIT Saline Indicator Method: A Self-Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EIT-BH-PERF-2025-01
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Lung Perfusion; Respiratory Physiology; Electrical Impedance Tomography; Ventilation-Perfusion Mismatch
Keywords: Electrical Impedance Tomography; Lung Perfusion; Saline Indicator; Breath-Hold; Inspiratory / Expiratory Phases; Regional Perfusion; Ventilation-Perfusion Matching
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Group - Self-Controlled (Experimental)
  Interventions: Procedure: Electrical Impedance Tomography Saline Indicator Procedure; Device: Electrical Impedance Tomography Device

INTERVENTIONS:
Procedure: Electrical Impedance Tomography Saline Indicator Procedure — Participants undergo continuous electrical impedance tomography (EIT) monitoring with a circumferential electrode belt placed around the thorax. During the procedure, participants perform standardized inspiratory and expiratory breath-hold maneuvers. At each breath-hold phase, a rapid intravenous bolus of sterile saline (10-20 mL) is administered, followed by a saline flush, to generate transient impedance changes for lung perfusion imaging using the saline indicator technique. EIT data are recorded continuously before, during, and after each saline injection. Each participant undergoes both breath-hold conditions and serves as their own control.
Device: Electrical Impedance Tomography Device — An FDA-cleared electrical impedance tomography (EIT) device is used to noninvasively monitor thoracic impedance changes during the study procedures. The device is used solely for physiological monitoring and image acquisition and is not being evaluated for safety, performance, or a new indication.

SUMMARY:
This study aims to compare lung perfusion distribution between inspiratory breath-hold and expiratory breath-hold phases using the saline indicator method combined with electrical impedance tomography (EIT). A self-controlled crossover design will be used in which each participant undergoes both breath-hold conditions with standardized rapid intravenous saline injections. The primary objective is to evaluate changes in global and regional pulmonary perfusion under different lung volume states. The findings may improve understanding of perfusion redistribution with lung inflation and support optimized ventilatory strategies in clinical practice.

DETAILED DESCRIPTION:
Electrical impedance tomography (EIT) with saline bolus injection is a noninvasive technique capable of generating real-time regional lung perfusion images based on transient impedance changes. Lung perfusion is highly dependent on lung volume, vascular resistance, and gravity, yet quantitative bedside evaluation remains limited.

This prospective self-controlled study investigates the differences in lung perfusion between inspiratory breath-hold (near total lung capacity) and expiratory breath-hold (near functional residual capacity). Each participant will undergo two standardized procedures: (1) expiratory breath-hold followed by a rapid intravenous injection of saline, and (2) inspiratory breath-hold followed by the same injection protocol. The order will be randomized.

Perfusion images will be reconstructed using time-impedance curves derived from saline indicator dilution. Regional perfusion parameters, including dependent vs nondependent zones and global perfusion distribution, will be compared between the two phases.

This study may provide foundational physiological evidence for understanding perfusion redistribution across lung volumes and support the clinical application of EIT in respiratory monitoring, ventilatory management, and rehabilitation in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Able to provide written informed consent
* Able to perform standardized inspiratory and expiratory breath-hold maneuvers for at least 8 seconds
* No known acute cardiopulmonary disease
* Suitable for noninvasive electrical impedance tomography monitoring and intravenous saline administration

Exclusion Criteria:

* Known severe cardiopulmonary disease (e.g., advanced chronic obstructive pulmonary disease, severe pulmonary hypertension, or heart failure)
* Hemodynamic instability or clinically significant cardiac arrhythmia
* Contraindication to intravenous saline administration or fluid bolus
* Pregnancy or breastfeeding
* Skin conditions or chest wall abnormalities preventing proper placement of EIT electrodes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Global Lung Perfusion Distribution | During the study procedure (within 1 hour)
  Quantitative assessment of global lung perfusion distribution derived from saline-induced impedance changes measured by electrical impedance tomography during inspiratory and expiratory breath-hold phases. Global perfusion is expressed as the percentage contribution of regional perfusion relative to total lung perfusion.

SECONDARY OUTCOMES:
Global Lung Perfusion Heterogeneity Index | During the study procedure (within 1 hour)
  Spatial heterogeneity of lung perfusion quantified using a perfusion heterogeneity index derived from regional perfusion maps obtained with the electrical impedance tomography saline indicator technique.